CLINICAL TRIAL: NCT02662361
Title: The Prevalence and Risk Factors for Patients With Peri-implant Disease：a Retrospective Study
Brief Title: Evaluation of the Prevalence and Risk Factors for Patients With Peri-implant Disease：a Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Ji-hua Chen, Professor and Dean of the Department of Prosthodontics, School of Stomatology, Fourth Military Medical University, Air Force Military Medical University, China
Other Study IDs: IRB-REV-2014027
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-01

CONDITIONS: Jaw, Edentulous, Partially
Keywords: peri-implant disease; risk factors; prevalence
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- no peri-implant disease: The subjects who did not suffer from peri-implant disease.
- peri-implant disease: The subjects who suffered from peri-implant disease.

SUMMARY:
To investigate the patient-related risk factors for peri-implant disease in partially edentulous patients rehabilitated with implants supported crown or bridge so as to provide evidence for clinical prevention and control.

DETAILED DESCRIPTION:
Objective: To investigate the patient-related risk factors for peri-implant disease in partially edentulous patients rehabilitated with implants supported crown or bridge so as to provide evidence for clinical prevention and control. Methods:A total of 131 patients will enroll in the study. Univariate and multivariate logistic regression analysis is used to determine the patient factors associated with peri-implant disease. The variables include age, gender, smoking and alcohol consumption, presence of diabetes, cardiovascular disease, osteoporosis, bruxism, bleeding upon brushing, reason for extraction, oral hygiene and periodontal status.

ELIGIBILITY:
Inclusion Criteria:

Patients implanted at least one implant and restored with implant-supported fixed partial dentures and single crowns.

The implant-supported fixed partial dentures and single crowns were in function at least one year.

Exclusion Criteria:

Jaw radiotherapy treatment before and after implanting. Patients who have bruxism, xerostomia or the adjacent teeth periapical periodontitis.

Patients who suffered with oral mucosa disease,or aggressive periodontitis or jaw defect.

Patients who suffered with mental and psychological disease will influence their oral health normal maintenance.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients restored with implant-supported fixed partial dentures and single crowns at the Department of Prosthodontics, School of Stomatology of the Fourth Military Medical University between January 2011 to May 2014.
Sampling Method: Probability Sample
Enrollment: 131 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Survival of implants | at the first return visit（at least one year after restoration）
  Time from the surgical placement of implants until the first return visit（at least one year after restoration）

SECONDARY OUTCOMES:
Gingival Bleeding on Probing | at the first return visit（at least one year after restoration）
  Gingival bleeding on probing (BOP) using the modified sulcus bleeding index for implants. Scale equals 0 = No bleeding when periodontal probe is passed along the gingival margin;1 = Isolated bleeding spots visible;2 = Blood forms a confluent red line on the gingival margin;3 = Heavy or profuse bleeding.
Pocket depths | at the first return visit（at least one year after restoration）
  Pocket depths measured around implants in millimeter (mm)
Marginal bone loss | at the first return visit（at least one year after restoration）
  Time from the surgical placement of implants until the first return visit（at least one year after restoration）

CONTACTS AND LOCATIONS:
Overall Officials: Yongjin Chen, 029-84776488, Principal Investigator — IRB of Stomatological Hospital of FMMU,PLA
Locations (1):
- Stomatological Hospital of Fourth Military Medical University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Ferreira SD, Silva GL, Cortelli JR, Costa JE, Costa FO. Prevalence and risk variables for peri-implant disease in Brazilian subjects. J Clin Periodontol. 2006 Dec;33(12):929-35. doi: 10.1111/j.1600-051X.2006.01001.x. PMID 17092244